CLINICAL TRIAL: NCT00761709
Title: Safety and Intraocular Pressure (IOP)-Lowering Efficacy of AL-39256 in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-08-28
Record Dates: First submitted 2008-09-25; First posted 2008-09-29 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- AL-39256 (Experimental): AL-39256 Ophthalmic Suspension, 1%, 1 drop in the study eye(s) at 8 AM from the morning bottle and 1 drop in the study eye(s) at 8 PM from the evening bottle for 4 weeks.
  Interventions: Drug: AL-39256 Ophthalmic Suspension, 1%
- XALATAN (Active Comparator): Latanoprost Ophthalmic Solution, 0.005%, 1 drop in the study eye(s) at 8 PM from the evening bottle (morning bottle contained vehicle and was dosed 1 drop in the study eye(s) at 8 AM) for 4 weeks.
  Interventions: Drug: Latanoprost Ophthalmic Solution, 0.005%; Drug: Vehicle
- Vehicle (Placebo Comparator): Inactive ingredients, 1 drop in the study eye(s) at 8 AM from the morning bottle and 1 drop in the study eye(s) at 8 PM from the evening bottle for 4 weeks.
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: AL-39256 Ophthalmic Suspension, 1%
  Arms: AL-39256
Drug: Latanoprost Ophthalmic Solution, 0.005%
  Other Names: XALATAN®
  Arms: XALATAN
Drug: Vehicle — Inactive ingredients used as a placebo comparator
  Arms: Vehicle; XALATAN

SUMMARY:
The purpose of this study is to evaluate the safety and intraocular pressure (IOP)-lowering efficacy of AL-39256 in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with open-angle glaucoma or ocular hypertension.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2009-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in IOP | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, Ph.D., Study Director — Alcon Research